CLINICAL TRIAL: NCT05275244
Title: PROSPECTIVE OBSERVATIONAL STUDY TO EVALUATE THE CLINICAL BENEFIT OF LOCAL TREATMENT WITH KD Intra-Articular® GEL (PRONOLIS® HD), IN PATIENTS WITH OSTEOARTHRITIS OF THE SHOULDER, HIP, ANKLE OR BASE OF THE THUMB
Brief Title: Evaluate Clinical Benefit of Local Treatment With KD Intra-Articular® Gel in Patients With Osteoarthritis (NO-DOLOR2)
Acronym: NO-DOLOR2
Status: Completed | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: NO-DOLOR-2-2021-02
Record Dates: First submitted 2022-02-10; First posted 2022-03-11 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis Thumb; Osteoarthritis Ankle
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteoarthritis Group: The patients diagnosed with single or preferential symptomatic osteoarthritis of the shoulder or hip treated with KD Intra-Articular® gel 2.2% - 44 mg in 2 ml - (Pronolis® HD one 2.2%), and ankle or base of the thumb treated with KD Intra-Articular® gel 1.6% - 16 mg in 1 ml - (Pronolis® HD mini 1.6%). Each patient will be administrated three injections, one per week.
  Interventions: Device: KD Intra-Articular® gel

INTERVENTIONS:
Device: KD Intra-Articular® gel — Depending on the joint, 3 injections will be administrated to the patient: KD Intra-Articular® gel 2.2% - 44 mg in 2 ml - (Pronolis® HD one 2.2%) in the case of shoulder and hip, or KD Intra-Articular® gel 1.6% - 16 mg in 1 ml - (Pronolis® HD mini 1.6%) in the case of the ankle and base of the thumb. The administration of the infiltrations will be with an interval of one week.

SUMMARY:
Prospective observational, national, multicentre, open study with a class III medical device with EC marking. Study to evaluate the clinical benefit of local treatment with KD intra-articular® gel in patients with osteoarthritis of the shoulder, hip, ankle or base of the thumb. The study will be conducted in the Rheumatology Service of Spanish Hospitals under the usual medical conditions, in accordance with routine clinical practice and following the internationally recognised precepts of good clinical practice of ICH and Declaration of Helsinki. The objective is to evaluate the evolution of pain in patients diagnosed with single or preferential symptomatic osteoarthritis of the shoulder or hip treated with KD Intra-Articular® gel 2.2% - 44 mg in 2 ml - (Pronolis® HD one 2.2%), and ankle or base of the thumb treated with KD Intra-Articular® gel 1.6% - 16 mg in 1 ml - (Pronolis® HD mini 1.6%).

Eighty patients will be included among about 6 Spanish Sites. The study comprises a maximum of 6 visits per protocol. At visit 0, informed consent will be obtained, the patient will be checked for fulfil the selection criteria. A pain assessment will also be carried out using a Visual Analogue Scale (VAS) and the corresponding questionnaire will be completed depending on the affected joint. According to the usual clinical practice of the site, the study treatment will be administered. A week after the first infiltration the second visit (V1) will be applied, and the VAS will be repeated. The patient's global clinical impression of change will also be assessed, and along with the Likert scale of satisfaction will be collected. The next visit (V2) will be carried out a week after the second infiltration and the procedures will be the same as those of the previous visit (V1). At 4 (V3), 12 (V4) and 24 (V5) weeks after receiving the third infiltration (V2), follow-up visits will be carried out where the assessment procedures will be the same as in visit 0, in addition to the GCI -C, the Likert scale of satisfaction and the collection of potential AEs and changes in concomitant medication. At each visit, the patient will be given a diary, where they will collect the rescue medication they have needed since the previous visit. In the electronic case report form (eCRF), the rescue medication (analgesics and NSAIDs) that you have needed since the previous visit (V0-V2) or in the month prior to the study visit (V3-V6) will be collected.

DETAILED DESCRIPTION:
Prospective observational, national, multicenter, open study with a class III medical device with EC marking. Study to evaluate the clinical benefit of local treatment with KD intra-articular® gel in patients with osteoarthritis of the shoulder, hip, ankle, or base of the thumb. The objective is to evaluate the clinical benefit of local treatment with KD Intra-Articular® gel 2.2% - 44 mg in 2 ml - (Pronolis® HD one 2, 2%), in patients with osteoarthritis of the shoulder or hip and with KD Intra-Articular® gel 1.6% - 16 mg in 1 ml - (Pronolis® HD mini 1.6%) in patients with osteoarthritis of the ankle or base of the thumb.

The study comprises a maximum of 6 visits per protocol. At visit 0, informed consent will be obtained, the patient will be checked for compliance with all inclusion criteria and no exclusion criteria in the study, and a medical history and physical examination will be carried out. A pain assessment will also be carried out using a VAS and the corresponding questionnaire will be completed depending on the joint to be treated (WOMAC, FAOS, ASES or DASH) and if it is the base of the thumb, the hand dynamometer test will be performed to obtain baseline results. According to the usual clinical practice of the center, the study treatment will be administered, or you will be summoned for administration at a later visit. A week after the first infiltration (V0) the second will be applied, and the VAS will be repeated (V1). The GCI-C evaluation by the patient and the Likert scale of satisfaction will also be carried out. AEs will be collected, if any, and if there have been changes in concomitant medication. The next visit (V2) will be carried out a week after the second infiltration has been placed and the procedures will be the same as those of the previous visit (V1). At 4 (V3), 12 (V4) and 24 (V5) weeks after receiving the third infiltration (V2), follow-up visits will be carried out where the assessment procedures will be the same as in visit 0, in addition to the GCI -C, the Likert scale of satisfaction and the collection of potential AEs and changes in concomitant medication.

At each visit, the patient will be given a diary, where they will collect the rescue medication they have needed since the previous visit. In the eCRF, the rescue medication (analgesics and NSAIDs) that you have needed since the previous visit (V0-V2) or in the month prior to the study visit (V3-V6) will be collected.

The study will be conducted under routine clinical practice conditions, with no restrictions being imposed on the participating doctor prescribing the drug(s) and no interference in normal clinical practice. Except for the scales and/or questionnaires used as measurement instruments in this study and a patient diary where the necessary rescue medication will be collected, the patients included will not be given any intervention, either diagnostic or follow-up, that is not the usual practice in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years.
2. Patients who come to a control consultation for single or preferential symptomatic osteoarthritis, primary in the case of the hip, shoulder or base of the thumb, or secondary post-traumatic in the case of the ankle.
3. Patients who meet the ACR diagnostic criteria for osteoarthritis of the hip and base of the thumb. Patients who meet the AOFAS diagnostic criteria for ankle osteoarthritis and those for shoulder osteoarthritis defined in the literature.
4. Patients with pain equal to or greater than 4 on the VAS pain scale.
5. Kellgren-Lawrence grade II-III patients in an X-ray performed within 18 months prior to inclusion.
6. Patients in whom viscosupplementation is indicated regardless of their inclusion in the study.
7. Patients able to read and understand the Patient Information Sheet and sign, if accepted, the Informed Consent Form.
8. Patients able, at the discretion of the investigator, to comply with the requirements of the study and without impediments to follow the instructions and assessments throughout the study.

Exclusion Criteria:

1. Known hypersensitivity to sodium hyaluronate or other study treatment components.
2. Previous trauma or surgical intervention in the affected joint (except in ankle osteoarthritis).
3. Participation in any other clinical trial or use of any drug or experimental device, currently or in the 4 weeks prior to inclusion in the study.
4. Swelling, exacerbation, or significant effusion in the affected joint.
5. Septic and aseptic arthritis.
6. Skin disorder or infection at the site of infiltration.
7. Patients requiring intra-articular infiltration in two joints.
8. Viscosupplementation of the affected joint within 6 months prior to the start of treatment.
9. Infiltration of steroids in the affected joint in the 3 months prior to the start of treatment.
10. History of autoimmune, microcrystalline rheumatological diseases or connective tissue diseases.
11. Coagulation disorders and/or anticoagulant medication that contraindicates infiltration.
12. Women who are pregnant, suspected of being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participation of 80 patients is expected (20 in each joint), diagnosed with osteoarthritis of the shoulder, hip, ankle or base of the thumb thanks to the collaboration of the rheumatology service of the public or private Spanish hospitals. The patients to be included in the study must meet all the above-mentioned screening criteria.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the evolution of the change in ankle osteoarthritis pain. | 24 weeks
  To evaluate the evolution of the change in ankle osteoarthritis pain, the Foot and Ankle Output Score (FAOS) questionnaire will be used. The mean questionnaire score at the 24-week visit versus baseline will be described.
To evaluate the evolution of the change in shoulder osteoarthritis pain. | 24 weeks
  To evaluate the evolution of the change in shoulder osteoarthritis pain, the American Shoulder and Elbow Surgeons (ASES) questionnaire will be used. The mean questionnaire score at the 24-week visit versus baseline will be described.
To evaluate the evolution of the change in pain in base of thumb. | 24 weeks
  To evaluate the evolution of the change in pain in base of thumb, the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used. The mean questionnaire score at the 24-week visit versus baseline will be described.
To evaluate the evolution of the change in hip osteoarthritis pain. | 24 weeks
  To evaluate the evolution of the change in pain in base of thumb, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire will be used. The mean questionnaire score at the 24-week visit versus baseline will be described.

SECONDARY OUTCOMES:
Assessment of the Need for Rescue Analgesic Medication. | 24 weeks
  To assess the change in the need for rescue analgesic medication at each follow-up visit vs. baseline visit, the percentage of patients who have increased/maintained/decreased the use of analgesics or NSAIDs with respect to the baseline visit.
Assessment of the Clinical Evolution by the Patient (1/2). | 24 weeks
  To assess the percentage of patients presenting improvement, > 20% improvement in the different domains of pain at the 24-week visits, the patients will be classified according to the percentage of improvement (relative change in the total score [if applicable] and in the scores of the domains other than pain) following the following cut-off points: > 0%, and > 20%. Additionally, these percentages of patients with improvement will be compared between both treatments.
Assessment of the Clinical Evolution by the Patient (2/2). | 24 weeks
  To assess the percentage of patients presenting improvement, > 50% improvement in the different domains of pain at the 24-week visits, the patients will be classified according to the percentage of improvement (relative change in the total score [if applicable] and in the scores of the domains other than pain) following the following cut-off points: > 0%, and > 50%. Additionally, these percentages of patients with improvement will be compared between both treatments.
Assessment of the Change in Grip Strength in Patients with Osteoarthritis of the Base of the Thumb. | 24 weeks
  To assess the evolution in grip strength, in patients with osteoarthritis of the base of the thumb, the mean test score obtained by the dynamometer at each follow-up visit will be described. In addition, the changes produced in this measurement between the 24-week visit and the baseline visit will be studied continuously (absolute change and relative change).
Evaluation of Patient Satisfaction with Treatment. | 24 weeks
  To assess the degree of patient satisfaction, the score obtained in the responses according to the Likert-type satisfaction scale at the 4-, 12- and 24-week visits will be described. Additionally, the results between both treatments will be compared.
Evaluation of Tolerability and Safety | 24 weeks
  To evaluate the tolerability of hyaluronic acid treatment, the percentage of patients who present AE to treatment during the observation period will be described, and a description of each of them will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991 May;34(5):505-14. doi: 10.1002/art.1780340502. PMID 2025304
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Gray R, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hand. Arthritis Rheum. 1990 Nov;33(11):1601-10. doi: 10.1002/art.1780331101. PMID 2242058
- [Background] Bryant D, Litchfield R, Sandow M, Gartsman GM, Guyatt G, Kirkley A. A comparison of pain, strength, range of motion, and functional outcomes after hemiarthroplasty and total shoulder arthroplasty in patients with osteoarthritis of the shoulder. A systematic review and meta-analysis. J Bone Joint Surg Am. 2005 Sep;87(9):1947-56. doi: 10.2106/JBJS.D.02854. PMID 16140808
- [Background] Domsic RT, Saltzman CL. Ankle osteoarthritis scale. Foot Ankle Int. 1998 Jul;19(7):466-71. doi: 10.1177/107110079801900708. PMID 9694125
- [Background] Lin W, Liu Z, Kampf N, Klein J. The Role of Hyaluronic Acid in Cartilage Boundary Lubrication. Cells. 2020 Jul 2;9(7):1606. doi: 10.3390/cells9071606. PMID 32630823